CLINICAL TRIAL: NCT01438632
Title: Pharmacology of Rapid-acting Insulin Injected by Needle-free Jet-injection in Patients With Diabetes
Brief Title: Pharmacology of Insulin Injected With Jet-injection in Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Pharma Group (EPG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PKPD_INSJ_2
Record Dates: First submitted 2011-09-19; First posted 2011-09-22 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus
Keywords: Insulin action; Jet injector; Diabetes Mellitus; Pharmacodynamics; Pharmacokinetics; Insulin analogs; Insulin aspart
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- jet injector (Experimental): Jet injectors deliver insulin at a high velocity (typically >100m/s) across the skin in the subcutaneous tissue, without the use of a needle
  Interventions: Device: jet injection device
- conventional insulin pen (Active Comparator)
  Interventions: Device: jet injection device

INTERVENTIONS:
Device: jet injection device — Rapid-acting insulin analogue aspart (Novorapid®) administration by means of a jet injector or a conventional insulin pen in the subcutaneous tissue. Dosage of insulin will be determined by the normal dosage of insulin used by the patient before breakfast.
  Other Names: Jet injector: InsuJet™ from the European Pharma Group; Insulin device: NovoPen® 3 from Novo Nordisk

SUMMARY:
A previous study showed that absorption and glucose-lowering action of rapid-acting insulin analogues occurred twice as fast when these analogues were administered by jet injection technology rather than by conventional insulin pen in healthy non-diabetic subjects. This study investigates if the rapid-acting insulin analogue aspart (Novorapid®) injected with jet-injection or a conventional insulin pen prior to a standardised meal in patients with diabetes shows the same difference in the pharmacokinetic and pharmacodynamic profile.

DETAILED DESCRIPTION:
A previous study showed that absorption and glucose-lowering action of rapid-acting insulin analogues occurred twice as fast when these analogues were administered by jet injection technology rather than by conventional insulin pen in healthy non-diabetic subjects. This study investigates if the rapid-acting insulin analogue aspart (Novorapid®) injected with jet-injection or a conventional insulin pen prior to a standardised meal in patients with diabetes (type 1 and type 2) shows the same difference in the pharmacokinetic and pharmacodynamic profile.The pharmacokinetic and pharmacodynamic profile of insulin aspart will be derived from the time-action profiles of insulin and glucose, respectively, in response to insulin injected directly prior to a standardised meal. All patients will be investigated twice, where on one occasion the jet-injector device will be used to inject an individualised dose of insulin and a conventional insulin pen to inject a placebo solution, and on the other occasion insulin will be injected with the conventional pen and placebo with the jet-injector. The order of these occasions will be randomised and blinded to both the investigator and the participating patient. The primary endpoint is the hyperglycaemic burden as reflected by area under the baseline-subtracted plasma glucose concentration time-curve from time 0 to 2 h after insulin injection and meal ingestion (BG-AUC0-2h). Secondary study endpoints are the area under the baseline-subtracted plasma glucose concentration time-curve from time 0 to 6 h (BG-AUC0-6h), maximal glucose excursion (BGmax), time to maximal glucose excursion (T-BGmax), time until plasma glucose has returned to baseline (T-BGBL), maximal insulin concentration (C-INSmax), time to maximal insulin concentration (T-INSmax), area under the insulin concentration curve (INSAUC) and time until 50% of insulin absorption (T-INSAUC50%) after insulin injection and meal ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Body-mass index 18-32 kg/m2
* Stable glycaemic control with HbA1c 6.0-9.0%
* Duration of diabetes >1 year
* Insulin use at least once daily or with subcutaneous pump
* Blood pressure <160/90 mmHg

Exclusion Criteria:

* Inability to provide informed consent
* Requirement of <8 units of rapid-acting insulin (analogue) before meals
* Chronic use of sulphonylurea derivatives, GLP-1 based treatments, acarbose or thiazolidinediones
* Treatment with prednisolone, non-steroidal anti-inflammatory drugs (NSAIDs), immunosuppressive agents, cytostatic drugs, hormone therapy except insulin, thyroid supplementation and oral anticonceptives
* Known allergy to aspart insulin
* Symptomatic diabetic neuropathy
* History of a major cardiovascular disease event (myocardial infarction, stroke, symptomatic peripheral artery disease, coronary bypass surgery, percutaneous coronary or peripheral artery angioplasty) in the past 6 months
* Pregnancy or the intention to become pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
BG-AUC0-2h (mmol•min-1•l-1): area under the baseline-subtracted plasma glucose concentration time-curve from time 0 to 2 h after insulin injection and meal ingestion. | 2 days (2 hours per day)
  based on plasma glucose levels during the first two hours of the 6-hour post-meal study duration

SECONDARY OUTCOMES:
BGmax (mmol/l): maximal glucose excursion after insulin injection and meal ingestion | 2 days (6 hours each day)
  Maximal plasma glucose value after the standardised meal
T-BGmax (min): time to maximal glucose excursion after insulin injection and meal ingestion | 2 days (6 hours per day)
  Time until maximal glucose value after the standardised meal and insulin injection
BG-AUC0-6h (mmol•min-1•l-1): area under the baseline-subtracted plasma glucose concentration time-curve from time 0 to 6 h after insulin injection and meal ingestion | 2 days (6 hours each day)
  Based on glucose concentration measurements for the total 6 hours of the study
T-BGBL (min): time until plasma glucose has returned to baseline values after insulin injection and meal ingestion | 2 days (6 hours per day)
  based on glucose level measurements during the total 6 hours of the study
T-INSmax (min): time to maximal insulin concentration (C-INSmax) | 2 days (6 hours per day)
  Maximal insulin concentration after insulin injection
INSAUC (pmol•min-1•l-1): area under the insulin concentration curve (from timepoint 0) | 2 days (6 hours per day)
  Based on insulin concentration measurements during the total 6 hours of the study
T-INSAUC50% (min): time until 50% of insulin absorption (mean residence time, MRT) | 2 days (6 hours each day)
  Based on insulin concentration measurements during the total 6 hours of the study
Number of patients requiring exogenous glucose infusion to prevent postprandial hypoglycaemia after insulin injection and meal ingestion | 2 days
  This will be assessed for the individual patient after every test. After completion of the experiments all cases of hypoglycemia will be assessed
Amount of exogenous glucose required to prevent postprandial hypoglycaemia after insulin injection and meal ingestion | 2 days
  This will be assessed for the individual patient after every test. After completion of the experiments the total amount of glucose infused will be calculate for each device
Duration of time that exogenous glucose is required to prevent postprandial hypoglycaemia after insulin injection and meal ingestion | 2 days
  This will be assessed for the individual patient after every test. After completion of the experiments the total amount of time will be calculate for each device
BG-AUC0-1h | 2 days (6 hours per day)
  the area under the baseline-subtracted plasma glucose concentration time-curve during the first hour

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan E de Galan, MD, PhD, Study Director — Radboud University Nijmegen Medical Centre, Department of general internal medicine 463, section Diabetes; Elsemiek EC Engwerda, BSc, Principal Investigator — Department of general internal medicine 463, section Diabetes, Radboud University Nijmegen Medical Centre
Locations (1):
- Department of general internal medicine 463, section Diabetes, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Mitragotri S. Current status and future prospects of needle-free liquid jet injectors. Nat Rev Drug Discov. 2006 Jul;5(7):543-8. doi: 10.1038/nrd2076. PMID 16816837
- [Background] Rave K, Klein O, Frick AD, Becker RH. Advantage of premeal-injected insulin glulisine compared with regular human insulin in subjects with type 1 diabetes. Diabetes Care. 2006 Aug;29(8):1812-7. doi: 10.2337/dc06-0383. PMID 16873785
- [Background] Engwerda EE, Abbink EJ, Tack CJ, de Galan BE. Improved pharmacokinetic and pharmacodynamic profile of rapid-acting insulin using needle-free jet injection technology. Diabetes Care. 2011 Aug;34(8):1804-8. doi: 10.2337/dc11-0182. Epub 2011 Jun 29. PMID 21715522